CLINICAL TRIAL: NCT01876745
Title: A Multicentre, Non-interventional, Observational Study to Evaluate Safety and Efficacy of NovoSeven® in Patients With Glanzmann's Thrombasthenia in Japan
Brief Title: A Study to Evaluate Safety and Efficacy of NovoSeven® in Patients With Glanzmann's Thrombasthenia in Japan
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-4030; U1111-1139-9589 (Other: WHO)
Record Dates: First submitted 2013-05-31; First posted 2013-06-13 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Congenital Bleeding Disorder; Glanzmann's Disease
MeSH Terms: conditions — Thrombasthenia | interventions — Factor VII; recombinant FVIIa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NovoSeven® (activated recombinant factor VII)
  Interventions: Drug: eptacog alfa (activated)

INTERVENTIONS:
Drug: eptacog alfa (activated) — Patients will be treated according to routine clinical practice at the direction of the treating physician. Data will be collected once a year after patient is registered with baseline visit until end of the study.
  Other Names: activated recombinant factor VII; NovoSeven®

SUMMARY:
This study is conducted in Asia. The aim of the study is to evaluate the safety and efficacy of NovoSeven® (activated recombinant factor VII, eptacog alfa (activated)) during bleeding episodes and for the prevention of bleeding during surgery/delivery in patients with Glanzmann's thrombasthenia (GT)/Glanzmann's disease.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities (Study related activity are any procedure related to recording of data according to the protocol).
* All-treated patients in the registration period

Exclusion Criteria:

* Known or suspected allergy to study product(s) or related products
* Septicaemia (especially, septicaemia followed severely infected patients caused by gram-negative bacteria [The risk of DIC (disseminated intravascular coagulation) caused by endotoxemia could not denied]
* Patients with a history of hypersensitivity to any of the product components

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with GT, who are enrolled in this study and to whom activated recombinant human factor VII (NovoSeven®) is administered in the study period, shall be included.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Therapy-related thrombosis | From onset of treatment until 6 hours after treatment onset

SECONDARY OUTCOMES:
Overall efficacy evaluated by the caregiver/patient: effective, partially effective, ineffective or not possible to evaluate | Within 30 days of end of treatment for bleeding episodes
Overall efficacy evaluated by the caregiver/patient: effective, partially effective, ineffective or not possible to evaluate | Within 24 hours after surgery for surgery/delivery

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com